CLINICAL TRIAL: NCT01688180
Title: The Prevalence and Impact of Depression and Anxiety Symptoms in Patients With Non-CF Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, yonghua gao, PHD, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: Yonghua Gao
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; depression; anxiety
MeSH Terms: conditions — Bronchiectasis; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with chronic diseases are at great risk of depression and anxiety.It is known that depression and anxiety are one of the most common comorbidities associated with chronic lung diseases such as asthma and chronic obstructive pulmonary disease.

However,to date,little is known about the rates and risk factors of depression and anxiety symptoms in non-CF bronchiectasis;and no large-scale prospective studies have been performed to investigate the effect of depression and anxiety on the healthy outcomes(such as number of exacerbations and hospitalizations over the ensuing year).Our purpose is to fill these gaps.

DETAILED DESCRIPTION:
Non-CF bronchiectasis is a long-term condition which affects the lungs.It is characterized by chronic airway infection with periodic exacerbations which are associated with impaired lung function, reduced quality of life and increased healthcare costs.Depression and anxiety are common and are known to be associated with poor quality of life and exacerbations of other chronic respiratory diseases such as COPD.Studies in COPD have shown that psychological distress is increasingly elevated and common,with up to 55% of patients suffering from a clinical diagnosis of anxiety and/or depression;moreover,patients with anxiety and/or depression were at greater risk for COPD-related exacerbations.Unfortunately,there has been no systematic evaluation of symptoms of depression and anxiety in patients with non-CF bronchiectasis or their relationship to health outcomes.A study including 111 non-CF bronchiectasis patients,O'Leary and colleagues indentified that 34% of patients had elevated scores for anxiety, depression or both.In a recent study of 93 patients(including 43 with Cystic fibrosis)of bronchiectasis,20% patients had elevated depression-related scores and 38 % had elevated anxiety-related scores,both depression and anxiety symptoms predicted signiﬁcantly worse health-related quality of life.

To date,the studies of depression and anxiety symptoms in patients with non-CF bronchiectasis have been limited by small samples sizes;and no prospective studies have been conducted to investigate the impact of psychological distress on the health outcomes.Given the importance of identifying and treating these symptoms, and their implications for long-term health outcomes,we plan to determine the prevalence and risk factors of depression and anxiety in non-CF bronchiectasis.In addition,we investigate the effect of depression and anxiety on the risk of non-CF bronchiectasis exacerbations and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. HRCT diagnosed Bronchiectasis
3. No fever,no worsening of respiratory symptoms,and no medication change within the 4 weeks before recruitment.
4. Capable of providing written informed consent

Exclusion Criteria:

1. cystic fibrosis
2. Previous lung transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with non-CF bronchiectasis attending the First Affiliated Hospital of Guangzhou Medical College,Guangzhou,Guangdong,China
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of depression and anxiety symptoms on non-CF bronchiectasis health outcomes. | one year
  Depression and anxiety are assessed at baseline using the Hospital Anxiety and Depression Scale(HADS).Health-related quality of life(HRQL) is measured using St.George's Respiratory Questionnaire(SGRQ), Leicester cough questionnaire(LCQ) and COPD assessment test(CAT) at baseline and follow-up.In the ensuing year,patients are monitored monthly by telephnone for 12 months to document the occurrence and characteristics of non-CF bronchiectasis exacerbations and hospitalizations.Patients are also encouraged to report to their investigators and research nurses whenever they experience symptom worsening.An exacerbation was defined as persistent (>24 hour) deterioration in at least three respiratory symptoms (including cough,dyspnoea, haemoptysis, increased sputum purulence or volume, and chest pain), with or without fever (>37.5˚ C),radiographic deterioration, systemic disturbances, or deterioration in chest signs.

SECONDARY OUTCOMES:
To estimate the prevalence of anxiety and depression symptoms in patients with non-CF bronchiectasis | six months
  Patients with non-CF bronchiectasis will complete the HADS, a brief, reliable and valid screening measure for depression and anxiety with well-established clinical cut-off scores.The HADS consists of seven items for depression(HAD-D) and seven items for anxiety(HAD-A).The scores range from 0 to 21 for each subscale,with a score of 0-7 denoting a noncase,8-10 a possible case,and 11 or higher a probable case.

OTHER OUTCOMES:
To identify risk factors associated with symptoms of depression and anxiety in patients with non-CF bronchiectasis | six months
  Demographic and clinical variables are collected ,including age,sex, body mass index(BMI),educational level,employment status,marital/partner status,amount of sputum produced daily,recent hemoptysis history,exacerbations in the previous year,6-minute walk test(6MWT),HRCT score,spirometry and sputum samples for microbiologic analysis at baseline.Some of these variables are collected again during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Chen, professor, Study Director — The First Affiliated Hospital of Guangzhou Medical University; Nanshan Zhong, Professor, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Gao YH, Guan WJ, Xu G, Gao Y, Lin ZY, Tang Y, Lin ZM, Li HM, Luo Q, Zhong NS, Birring SS, Chen RC. Validation of the Mandarin Chinese version of the Leicester Cough Questionnaire in bronchiectasis. Int J Tuberc Lung Dis. 2014 Dec;18(12):1431-7. doi: 10.5588/ijtld.14.0195. PMID 25517807